CLINICAL TRIAL: NCT04854512
Title: Randomized, Multicenter, Double-blind, Parallel-Group, Placebo & Comparator-Controlled Study to Compare the Glycemic Effects, Safety & Tolerability of Metformin Delayed-Release Tablets in Patients With Type 2 Diabetes Mellitus
Brief Title: Investigational Study of Delayed Release Metformin
Acronym: DREAM-T2D
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic company decision - not related to a safety concern
Sponsor: Anji Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANJ900D3501
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Investigational Arm (Metformin DR plus metformin IR placebo) (Experimental): Group A will receive 1800 mg Metformin DR qAM + placebo for 1500 mg metformin IR in divided doses (2×placebo for metformin IR 500 mg qAM and 1×placebo for metformin IR 500 mg qPM).
  Interventions: Drug: Metformin DR; Drug: Metformin IR placebo
- Placebo Arm (Metformin DR placebo plus metformin IR placebo) (Placebo Comparator): Group B will receive placebo for 1800 mg Metformin DR qAM + placebo for 1500 mg metformin IR in divided doses (2× placebo for metformin IR 500 mg qAM and 1×placebo for metformin IR 500 mg qPM).
  Interventions: Drug: Metformin DR Placebo; Drug: Metformin IR placebo
- Active Control Arm (Metformin DR placebo plus metformin IR) (Active Comparator): Group C will receive placebo for 1800 mg Metformin DR qAM + 1500 mg metformin IR in divided doses (2× metformin IR 500 mg qAM and 1× metformin IR 500 mg qPM).
  Interventions: Drug: Metformin IR; Drug: Metformin DR Placebo

INTERVENTIONS:
Drug: Metformin DR — Delay-Release Metformin
  Other Names: ANJ900; MetDR
  Arms: Investigational Arm (Metformin DR plus metformin IR placebo)
Drug: Metformin IR — Immediate Release Metformin
  Arms: Active Control Arm (Metformin DR placebo plus metformin IR)
Drug: Metformin DR Placebo — Metformin DR Placebo
  Arms: Active Control Arm (Metformin DR placebo plus metformin IR); Placebo Arm (Metformin DR placebo plus metformin IR placebo)
Drug: Metformin IR placebo — Metformin IR placebo
  Arms: Investigational Arm (Metformin DR plus metformin IR placebo); Placebo Arm (Metformin DR placebo plus metformin IR placebo)

SUMMARY:
In Phase 1 and 2 studies already conducted, Metformin DR, with its targeted delivery to the distal small intestine, has shown the potential to be a safe and effective way to improve glycemic control in patients with T2DM and CKD with less systemic metformin exposure. The primary purpose of this Phase 3 clinical study is to collect pivotal data confirming the safety and efficacy of Metformin DR in T2DM patients with varying renal function from normal up to CKD3B.

DETAILED DESCRIPTION:
The study is a multicenter, international study with a 28 week randomized, double blind parallel group, placebo and active comparator controlled period and a 24 week open label extension period in patients with T2DM who are treated with metformin at the time of study screening.

Approximately 675 patients will be randomly assigned to 1 of 3 treatment groups. The study will assess change in HbA1c through 28 weeks for Metformin DR compared to placebo as a primary endpoint. In addition, assessments of change in HbA1c for Metformin DR compared to Metformin IR and assessment of absolute change in HbA1c will be evaluated in the study.

Screening and Run-in Period:

The study will include an up to 10-day screening period, an 4 to 8-week metformin washout period, and a 2-week single blind (patient blinded) placebo run-in period.

Treatment Period:

Patients that are determined eligible based upon the screening and run-in criteria will enter the 28-week double-blind treatment period. During the double-blind treatment period, patients will be randomly assigned to 1 of 3 treatment groups (Group A, B, or C) in a 1:1:1 ratio. The 3 treatments are Metformin DR (1800 mg Metformin DR with matching placebo for Metformin IR), Metformin IR (1500 mg Metformin IR with matching placebo for Metformin DR), and placebo (matching placebo for Metformin IR with matching placebo for Metformin DR). For those patients randomized to Metformin IR, their Metformin IR dose will be titrated to prevent gastrointestinal intolerability:

Open Label Extension Period:

Upon completion of the 28 week treatment patients will be eligible for an additional 24 weeks of open label extension period where assigned study treatment will continue and additional efficacy, safety and tolerability data will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female and at least 18 years old
2. Has body mass index 20.0 to 45.0 kg/m2 (inclusive)
3. Has T2DM
4. Has HbA1c of 7.0% to 9.5%, inclusive, at Visit 1A and HbA1c value of 7.0% to 10.5%, inclusive, at Week -2 (Visit 3/3A as applicable)
5. Has an eGFR value of ≥30 mL/min/1.73 m2 based on the CKD-EPI equation at Visit 1A and Visit 3/3A (Week -2)
6. Stable treatment with a metformin preparation or a combination product containing metformin for 8 weeks prior to Visit 1A
7. If treated with the following medications, must be on a stable regimen for a minimum of 6 weeks prior to Visit 1B

   1. Drugs known to affect body weight, including prescription medications (e.g., phentermine, phentermine/topiramate, orlistat, lorcaserin, bupropion/naltrexone) and over-the-counter anti-obesity agents
   2. Hormone replacement therapy (female patients) and testosterone (male patients)
   3. Oral contraceptives (female patients)
   4. Antihypertensive agents including ACEi/ARB
   5. Lipid-lowering agents
   6. Thyroid replacement therapy
   7. Antidepressant agents
8. Ability to understand and willingness to adhere to protocol requirements

Exclusion Criteria:

1. Is currently on dialysis, has been on any dialysis within 1 year of Visit 1B, or is expected to undergo dialysis during the study period
2. Has a history of lactic acidosis
3. Has a fasting plasma glucose (FPG) value >240 mg/dL (>13.3 mmol/L) at Week -2 (Visit 3/3A as applicable)
4. An alanine aminotransferase or aspartate aminotransferase result >2.5 × upper limit of normal (ULN) or a bilirubin result >1.5 × ULN at Visit 1B or Visit 3/3A (Week -2) (except in case of documented Gilbert's syndrome)
5. Has a fasting plasma lactate value >2 mol at Visit 1B
6. Has a bicarbonate value ≤20 mEq/L at both Visit 1A and 1B. If bicarbonate value is <20 at Visit 3/3A or 4, patient may be excluded if the investigator considers this clinically significant
7. A history of >5% weight change within 12 weeks prior to Visit 1A
8. Has mean BP measurements >180 mmHg (systolic BP) or >100 mmHg (diastolic BP) at Visit 1A or Visit 3/3A, which can be rechecked within 1 week (Note: re-screening is allowed 6 weeks after initiation/modification of antihypertensive agents if the patient is screen failed due to BP only)
9. Oral antidiabetic agent or insulin use that is not stable for 8 weeks prior to randomization (i.e., change in oral medication dose or basal insulin dose increased or decreased by more than 20% during the 8 weeks prior to Visit 4 [Day 1])
10. Has been treated, is currently being treated, or is expected to require or undergo treatment with any of the following excluded medications:

    1. Prescribed metformin preparation after initiation of metformin washout following Visit 1B
    2. Greater than 10 consecutive days of systemic corticosteroids by oral, intravenous, or intramuscular route within 12 weeks of Visit 1B; inhaled, intranasal, ophthalmic, topical, or intra-articular corticosteroids are not exclusionary
    3. Planned use of proton pump inhibitors after Visit 2 (Week -6); such use could potentially affect the DR and PK of Metformin DR. Proton pump inhibitor treatment may be replaced by other treatment (such as H2 receptor antagonists [excluding ranitidine], or calcium carbonate antacids) prior to Visit 4 (Day 1), if appropriate per the judgment of the Investigator
    4. Cationic drugs that are eliminated by renal tubular secretion (e.g., amiloride, digoxin, morphine, procainamide, flecainide, quinidine, quinine, ranitidine, triamterene, trimethoprim, and vancomycin) within 1 week of Visit 3 (Week 2)
    5. Iodinated contrast dye within 1 week prior to Visit 3 (Week -2)
    6. Investigational drug within 8 weeks (or 5 half-lives of the investigational drug, whichever is greater) of the date of the first dose of randomized study medication
    7. Metformin DR or double-blind matching placebo for Metformin DR at any time prior to Visit 1B
11. Has a clinically significant medical condition as judged by the Investigator that could potentially affect study participation and/or personal well-being, including but not limited to the following conditions:

    1. Hepatic disease
    2. Gastrointestinal disease, including but not limited to:

    i. History or presence of inflammatory bowel disease or other severe gastrointestinal disease, particularly those that may impact gastric emptying, such as gastroparesis and pyloric stenosis ii. Prior or expected surgical gastrointestinal procedure that may impact the gut hormonal response to study medication such as gastric bypass surgery or gastric banding surgery iii. Active diagnosis of pancreatitis c. Endocrine disorder other than T2DM or hypothyroidism on replacement therapy d. Cardiovascular disease, including history of stroke, decompensated heart failure New York Heart Association Class III or IV, myocardial infarction, unstable angina pectoris, or coronary arterial bypass graft or angioplasty within 3 months prior to Visit 1A (screening) e. Central nervous system diseases such as epilepsy f. Psychiatric or neurological disorders that in the Investigator's opinion would cause the patient to be noncompliant with study procedures g. Organ transplantation h. Chronic or acute infection requiring systemic antibiotic treatment i. Orthostatic hypotension or syncope j. Active malignancy within the past 5 years with exception of basal cell and squamous cell carcinoma
12. Known allergy or hypersensitivity to Metformin DR, Metformin IR, or placebo or any inactive component of study medication, active comparator, or placebo, unless the reaction is deemed irrelevant to the study by the Investigator (prior history of gastrointestinal intolerance to metformin is not exclusionary)
13. Has a history of diabetic ketoacidosis or hyperosmolar non-ketotic hyperglycemia within 1 year prior to Visit 1B
14. A physical, psychological, or historical finding that, in the Investigator's opinion, would make the patient unsuitable for the study
15. Any verified clinically significant abnormality identified on physical examination, laboratory tests, ECG, vital signs, or any adverse event (AE) at the time of Visit 1B through Visit 4 that, in the judgment of the Investigator or any Sub-investigator, would preclude safe completion of the study or constrains efficacy assessment
16. Currently abuses drugs or alcohol or has a known history of abuse that in the Investigator's opinion would cause the patient to be noncompliant with study procedures
17. Had a blood transfusion or experienced significant blood loss (i.e., >500 mL), including loss due to blood donation, within 8 weeks prior to Visit 1B, or is planning to donate blood or have a blood transfusion during the study
18. Prior or planned major surgery of any kind (requiring overnight hospitalization) within 6 months of Visit 1B
19. Patients insufficiently compliant with study medication during the placebo run-in phase (<85% or >115%) as assessed at Visit 4
20. Is screening for the study at more than one clinical site or is participating in any other clinical study
21. Is currently pregnant (confirmed by serum pregnancy test at Visit 1B) or breastfeeding or plans to become pregnant during the course of the study
22. Women of childbearing potential not willing to use highly effective method(s) of birth control during the entire study, or who are unwilling or unable to be tested for pregnancy
23. If the patient has evidence of coronavirus disease 2019 (COVID-19) within 2 weeks prior to enrolment (a positive COVID-19 test or suspicion of COVID-19 infection), the patient cannot be enrolled in the study
24. Is employed by Anji Pharma (that is an employee, contract worker, or designee of the company).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 675 (Estimated)
Dates: Start 2021-05-18 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | Baseline to 28 weeks
  Change in HbA1c in patients treated with Metformin DR compared to placebo

SECONDARY OUTCOMES:
HbA1c response (Metformin DR vs. placebo) | Baseline to 28 weeks
  HbA1c absolute value-based response (Yes/No) at Week 28 defined as HbA1c ≤7% for Metformin DR compared to placebo
Change in HbA1c (Met DR vs. metformin IR) | Baseline to 28 weeks
  Change in HbA1c from the double-blind treatment period baseline to Week 28 for Metformin DR compared to Metformin IR
HbA1c response (Metformin DR vs. metformin IR) | Baseline to 28 weeks
  HbA1c absolute value-based response (Yes/No) at Week 28 defined as HbA1c ≤7% for Metformin DR compared to Metformin IR.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Meyers, MD, Study Chair — Chief Medical Officer - Anji Pharma
Locations (87):
- United States (33):
  - Lenzmeier Family Medicine/CCT Research, Glendale, Arizona
  - Aventiv Research, Mesa, Arizona
  - Kidney & Hypertension Center / DaVita Clinical Research, Apple Valley, California
  - California Institute of Renal Research, Chula Vista, California
  - Academic Medical Research Institute, Los Angeles, California
  - Valley Renal Medical Group Research, Northridge, California
  - San Fernando Valley Health Institute, Van Nuys, California
  - AGA Clinical Trials, Hialeah, Florida
  - East Coast Institutue for Research, Jacksonville, Florida
  - East Coast Institute for Research, LLC, Lake City, Florida
  - West Orange Endocrinology, Ocoee, Florida
  - Metabolic Research Institute, Inc, West Palm Beach, Florida
  - Georgia Nephrology Research Institute, Lawrenceville, Georgia
  - In-Quest Medical Research - Peachtree, Peachtree Corners, Georgia
  - Louisville Metabolic and Atherosclerosis Research Center Inc. (L-MARC), Louisville, Kentucky
  - Methodist Physicians Clinic / CCT Research, Fremont, Nebraska
  - Midwest Regional Health Services, Omaha, Nebraska
  - DaVita Clinical Research, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Carolina Institute for Clinical Research, Fayetteville, North Carolina
  - Lucas Research, Morehead City, North Carolina
  - Eastern Nephrology Associates, New Bern, North Carolina
  - Family Medicine of SayeBrook, Myrtle Beach, South Carolina
  - South Carolina Clinical Research LLC, Orangeburg, South Carolina
  - WR-ClinSearch, Chattanooga, Tennessee
  - Texas Diabetes & Endocrinology, Austin, Texas
  - Office of Osvaldo A Brusco, MD, Corpus Christi, Texas
  - Galenos Research, Dallas, Texas
  - Endocrine IPS, PLLC, Houston, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas
  - Manassas Clinical Research Center, Manassas, Virginia
  - IACT Health, Suffolk, Virginia
- Brazil (10):
  - Instituto de Ensino e Pesquisa Clinica do Ceara, Fortaleza, Ceará
  - Centro de Pesquisas em Diabetes e Doencas Endrocrino-Metabolica Ltda, Fortaleza, Ceará
  - Centro de Diabetes Curitiba, Curitiba, Paraná
  - Cline Research Center, Curitiba, Paraná
  - Universidade Federal Do Para (UFPA) - Insitituto de Ciencas de Saude (ICS), Belém, Pará
  - IBPClin Instituto Brasil de Pesquisa Clinica, Rio de Janeiro, Rio de Janeiro
  - Hospital Sao Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Centro de Pesquisas em Diabetes Ltda, Porto Alegre, Rio Grande do Sul
  - Loema - Instituto de Pesquisa Clinica, Campinas, São Paulo
  - Instituto de Pesquisa Clinica de Campinas, Campinas, São Paulo
- Bulgaria (7):
  - ASOMC Endocrinology and Metabolic Diseases, Rousse
  - Medical Cetner Teodora, Rousse
  - Multiprofile Hospital for Active Treatment, Smolyan
  - Fourth Multipfoile Hospital for Active Treatment, Sofia
  - Medical Center New Rehabilition Cetner EOOD, Stara Zagora
  - Diagnostic Culsultative Cetner "Equita" EOOD, Varna
  - Medical Center Leo Clinical EOOD, Varna
- Canada (8):
  - BC Diabetes, Vancouver, British Columbia
  - LMC Manna Research (Barrie), Barrie, Ontario
  - LMC Manna Research (Brampton), Brampton, Ontario
  - Stephen S. Chow Medicine Professional Corporation, East York, Ontario
  - LMC Manna Research (Etobicoke), Etobicoke, Ontario
  - LMC Manna Research (Ottawa), Nepean, Ontario
  - LMC Manna Research (Bayview), Toronto, Ontario
  - LMC Manna Research (Montreal), Montreal, Quebec
- Czechia (7):
  - Diahaza s.r.o., Holešov
  - Diabetologicka ambulance, Krnov
  - Interni Ambulance, Olomouc
  - Endodiab s.r.o., Prague
  - Diabet2 s.r.o., Prague
  - Diabetologicka a podiatricka ambulance, Milan Kvapil s.r.o., Prague
  - ResTrial s.r.o., Prague
- Hungary (8):
  - Borbanya Praxis EU Kft, Nyíregyháza, SZ
  - Lausmed Kft, Baja
  - Principal SMO Ltd, Baja
  - DRC Gyogyszervizsgalo Kozpont Kft, Balatonfüred
  - Bajscy-Zsilinszky Hospital, Budapest
  - Magyar Honvedseg Egeszsegugyl Koxpont, Budapest
  - Borbanya Praxis EU k ft, Debrecen
  - Zala Megyei Szent Rafael Korhaz, Zalaegerszeg
- Poland (9):
  - Malopolskie Centrum Kliniczne, Krakow, Lesser Poland Voivodeship
  - NZOZ NEUROMED M.iM. Nastaj Sp.P., Lublin, Lublin Voivodeship
  - Niepubliczny Zakład Opieki Zdrowotnej Specjalistyczny Ośrodek Internistyczno-Diabetologiczny, Bialystok
  - Centrum Medyczne Pratia, Katowice
  - Pro Familia Altera Sp. z.o.o., Katowice
  - Diamond Medical Center, Krakow
  - NBR Polska, Warsaw
  - Centralny Szpital Kliniczny Ministerstwa Spraw Wewnetrznych i Administracji, Warsaw
  - Centrum Badan Klinicznych Piotr Napora Lekarze Spolka Partnerska, Centrum Badan Klinicznych Osrodek Badan Wczesnej Fazy, Wroclaw
- Spain (5):
  - Hospital Universitario Virgen del Rocio, Seville, SE
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Nuevas Tecnologias en Diabetes y Endocrinologia, Seville
  - Hospital Vithas Sevilla, Seville

IPD SHARING:
Plan to Share IPD: No